CLINICAL TRIAL: NCT00862524
Title: A Study of ARRY-334543 and Gemcitabine in Patients With Advanced Cancer and Pancreatic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Array BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARRAY-543-206
Record Dates: First submitted 2009-03-16; First posted 2009-03-17 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-09

CONDITIONS: Advanced Cancer; Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — ARRY-334543; Gemcitabine; Nucleosides

ARMS (1):
- ARRY-334543 + gemcitabine (Experimental)
  Interventions: Drug: ARRY-334543, EGFR/ErbB2 inhibitor; oral; Drug: Gemcitabine, nucleoside analogue; intravenous

INTERVENTIONS:
Drug: ARRY-334543, EGFR/ErbB2 inhibitor; oral — multiple dose, escalating
Drug: Gemcitabine, nucleoside analogue; intravenous — multiple dose, single schedule

SUMMARY:
This is a 2-phase study during which patients with advanced/metastatic solid tumors will receive investigational study drug ARRY-334543 and gemcitabine.

The study has 2 parts. In the first part of the study, Phase 1, patients with advanced/metastatic solid tumors will receive increasing doses of study drug in combination with gemcitabine in order to achieve the highest dose of study drug possible that will not cause unacceptable side effects. Patients will be followed to see what side effects the combination causes and what effectiveness the combination has, if any, in treating the cancer. Approximately 24 patients from the US will be enrolled in Part 1 (Completed).

In the second part of the study, Phase 2, patients with metastatic pancreatic cancer will receive the best dose of study drug, in combination with gemcitabine, determined from the first part of the study and will be followed to see what side effects the combination causes and what effectiveness the combination has, if any, in treating the cancer. Approximately 42 patients from the US will be enrolled in Part 2 (Withdrawn).

ELIGIBILITY:
Key Inclusion Criteria (Part 1):

* Histologically or cytologically confirmed diagnosis of a solid tumor suitable for treatment with gemcitabine.
* No more than 3 prior anticancer regimens for advanced disease.
* Measurable or evaluable, nonmeasurable disease.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1.
* Able to take and retain oral medications.
* Additional criteria exist.

Key Exclusion Criteria (Part 1):

* Uncontrolled or symptomatic brain metastases (if a patient has brain metastases and is on steroids, the steroid dose must have been stable for at least 30 days).
* Treatment with prior chemotherapy within 21 days of first dose of study drug.
* Requiring IV alimentation.
* Pregnancy or lactation.
* Known positive serology for the human immunodeficiency virus (HIV), hepatitis B and/or hepatitis C.
* History of being unable to tolerate gemcitabine or any of its components.
* Additional criteria exist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-03; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Establish the maximum tolerated dose (MTD) of study drug in combination with gemcitabine. | Part 1
Characterize the safety profile of study drug in combination with gemcitabine in terms of adverse events, clinical laboratory tests and electrocardiograms. | Part 1
Characterize the pharmacokinetics (PK) of study drug, gemcitabine and a gemcitabine metabolite. | Part 1
Assess the efficacy of the study drug in combination with gemcitabine in terms of progression-free survival (PFS) at 16 weeks. | Part 2

SECONDARY OUTCOMES:
Assess the efficacy of the study drug in combination with gemcitabine in terms of tumor response. | Part 1
Characterize the safety profile of study drug in combination with gemcitabine in terms of adverse events, clinical laboratory tests and electrocardiograms. | Part 2

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Pinnacle Oncology/Hematology, Phoenix, Arizona
  - Premiere Oncology, Santa Monica, California
  - University of Colorado Health Sciences Center, Aurora, Colorado
  - Partners, Massachusetts General Hospital, Boston, Massachusetts
  - Partners, Dana Farber, Boston, Massachusetts
  - Sarah Cannon Research Center, Nashville, Tennessee